CLINICAL TRIAL: NCT00735462
Title: A Safety and Effectiveness Study of Imiquimod Creams in the Treatment of External Genital Warts
Brief Title: Phase 3 Study of Imiquimod Creams in the Treatment of External Genital Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Jason Wu, MD / Executive Director, Product Development, Graceway Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW01-0805
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-06

CONDITIONS: Genital Warts
Keywords: external genital warts; perianal warts; condylomata acuminata; human papilloma virus; HPV types 6 and 11
MeSH Terms: conditions — Condylomata Acuminata

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2.5% imiquimod cream (Experimental): 2.5% imiquimod cream applied daily to wart areas for up to 8 weeks
  Interventions: Drug: 2.5% imiquimod cream
- 3.75% imiquimod cream (Experimental): 3.75% imiquimod cream applied daily to wart areas for up to 8 weeks.
  Interventions: Drug: 3.75% imiquimod cream
- Placebo cream (Placebo Comparator): Placebo cream applied daily to wart areas for up to 8 weeks.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: 2.5% imiquimod cream — 2.5% imiquimod cream applied daily to wart areas for up to 8 weeks.
  Other Names: 2.5% imiquimod topical cream
  Arms: 2.5% imiquimod cream
Drug: 3.75% imiquimod cream — 3.75% imiquimod cream applied daily to wart areas for up to 8 weeks
  Other Names: 3.75% imiquimod topical cream
  Arms: 3.75% imiquimod cream
Drug: Placebo cream — Placebo cream applied daily to wart areas for up to 8 weeks
  Other Names: Placebo topical cream
  Arms: Placebo cream

SUMMARY:
The purpose of this study is to determine whether imiquimod creams are effective in treating external genital warts (EGW). The secondary objective of this study is to provide information on recurrence of EGW. Additionally the study will also look at any adverse events associated with the use of the creams.

External genital and perianal warts are caused by the infection of human papillomavirus or HPV. HPV infection is a sexually transmitted disease (STD). External genital warts look like small flesh-colored, pink, or red growths on or around the external skin of sex organs or perianal area. The warts may look similar to the small parts of a cauliflower or they may be very tiny and difficult to see. They often appear in clusters of three or four, and may grow and spread rapidly. They usually are not painful, although they may cause mild pain, bleeding, and itching.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Diagnosis of external genital / perianal warts with at least 2 warts and no more than 30 warts
* Negative pregnancy test (for women who are able to become pregnant)

Exclusion Criteria:

* Women who are pregnant, lactating or planning to become pregnant during the study
* Evidence of clinically significant or unstable disease (such as stroke, heart attack)
* Have any of the following conditions: HIV infection; current or history of high risk HPV infection (e.g., HPV types 16, 18, etc.); outbreak of herpes genitalia in the wart areas; internal warts requiring or undergoing treatment; dermatological disease (e.g., psoriasis) or skin condition in the wart areas
* Have received specific treatments in the treatment area(s) within the designated time period prior to study treatment initiation

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2008-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, MD, Study Director — Graceway Pharmaceuticals
Locations (43):
- United States (43):
  - NEA Clinic, Jonesboro, Arkansas
  - Northern Claifornia Research, Carmichael, California
  - California State University - Chico, Chico, California
  - Dermatology Research Associates, Los Angeles, California
  - Conant Foundation, San Francisco, California
  - Downtown Women's Healthcare, Denver, Colorado
  - Altus Research, Lake Worth, Florida
  - PMI Health Research Group, Atlanta, Georgia
  - Atlanta Women's Research Institute, Atlanta, Georgia
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Howard Brown, Chicago, Illinois
  - Valley Medical Center, Flint, Michigan
  - Women's OB/GYN, Saginaw, Michigan
  - Clayton Research Institute, St Louis, Missouri
  - Women's Health Research Center, Lawrenceville, New Jersey
  - Alliance Women's Research, Riverside Park, New Jersey
  - Southwest Clinical Research, Albuquerque, New Mexico
  - University Urology Associates, New York, New York
  - Boro Park ObGyn, New York, New York
  - Crescent Medical Research, Salisbury, North Carolina
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Rapid Medical Research, Cleveland, Ohio
  - Complete Healthcare for Women, Columbus, Ohio
  - Wright State University, Dayton, Ohio
  - Heartland Health Institute, Tulsa, Oklahoma
  - Clinical Trials of America, Eugene, Oregon
  - Westover Heights Clinic, Portland, Oregon
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Palmetto Clinical Research, Greer, South Carolina
  - Alpha Clinical Research, Clarksville, Tennessee
  - Adams Patterson Gynecology and Obstetrics, Memphis, Tennessee
  - Tennessee Women's Care, Nashville, Tennessee
  - DiscoveResearch, Bryan, Texas
  - TMC Life Research, Houston, Texas
  - West Houston Clinical Research Services, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - The Center for Clinical Studies, Webster, Texas
  - Utah Clinical Trials, Salt Lake City, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - CARE-ID, Annandale, Virginia
  - Tidewater Clinical Reseach, Virginia Beach, Virginia
  - Independence Family Medicine Clinical Research, Virginia Beach, Virginia
  - Women's Clinical Research Center, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.5% Imiquimod Cream: 2.5% imiquimod cream applied once daily to wart areas for up to 8 weeks.
- 3.75% Imiquimod Cream: 3.75% imiquimod cream applied once daily to wart areas for up to 8 weeks.
- Placebo: Placebo cream applied once daily to wart areas for up to 8 weeks.
Period: Overall Study
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Started | 202 | 204 | 105
Completed | 139 | 149 | 77
Not Completed | 63 | 55 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo | Total
Number analyzed (Participants) | 202 | 204 | 105 | 511
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 0 | 3
  Between 18 and 65 years | 201 | 201 | 104 | 506
  >=65 years | 0 | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 33.1 (10.1) | 32.8 (11.0) | 33.3 (10.8) | 33.1 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 116 | 56 | 289
  Male | 85 | 88 | 49 | 222
Region of Enrollment [Number; unit: participants]
  United States | 202 | 204 | 105 | 511

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Complete Clearance of All Warts (Baseline and New) at the End of Study.
Description: The complete clearance was defined as completely cleared all warts including baseline and newly emerged during the study at all anatomic areas.
Time Frame: Up to 16 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Number analyzed (Participants) | 202 | 204 | 105
proportion of participants | 0.248 [0.190 to 0.313] | 0.294 [0.233 to 0.362] | 0.09 [0.040 to 0.156]

2. Secondary Outcome: Number of Subjects With Any Treatment Related Adverse Reactions (AEs), Any Local Skin Reactions (LSRs), and Number of Subjects Who Took Rest Periods During the Treatment Period
Description: Treatment related defined as "probably related" or "related" by investigator. Local skin reactions (LSRs)were part of the treatment related adverse events and assessed by the investigators.
  Rest periods defined as temporary interruption of dosing due to intolerable local skin reaction.
Time Frame: Up to 16 weeks
Population: Analysis population was based on safety population which defined as for all subjects randomized and received at lease one dose. There was one subject who randomized to the 2.5% group but received one treatment kit of 3.75% imiq cream, so this subject was assigned to 3.75% for the safety analysis.
Measure: Number; unit: participants
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Number analyzed (Participants) | 201 | 205 | 105
participants
  Subjects with and Adverse Reactions (ARs) | 37 | 40 | 3
  Subjects with Any Local Skin Reactions (LSRs) | 123 | 148 | 41
  Number of Subjects who Took a Rest Period | 55 | 67 | 3

ADVERSE EVENTS:
Time Frame: One year
Description: The study period included 4 month enrollment, maximum 28 weeks of study phase, so total length of the study from first patient enrolled to last patient completed the study is about 11 months.
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Serious Adverse Events (participants affected / at risk) | 2/201 | 6/205 | 1/105
Other Adverse Events (participants affected / at risk) | 37/201 | 40/205 | 3/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5% Imiquimod Cream (N=201) | 3.75% Imiquimod Cream (N=205) | Placebo (N=105)
Malignant melanoma (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cystectomy (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5% Imiquimod Cream (N=201) | 3.75% Imiquimod Cream (N=205) | Placebo (N=105)
Application site pain (General disorders) | 8 (8) | 16 (16) | 0 (0)
Application site pruritus (General disorders) | 14 (14) | 7 (7) | 1 (1)
Application site irritation (General disorders) | 8 (8) | 11 (11) | 1 (1)
Application site rash (General disorders) | 3 (3) | 2 (2) | 0 (0)
Application site ulcer (General disorders) | 3 (3) | 2 (2) | 0 (0)
Application site bleeding (General disorders) | 1 (1) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
There was a high percentage of lost to follow up in this study. Since the disease studied in this study can be wait and watch, typically a high lost to follow up rate were seen in these kind of trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
a term restricts that PI can publish their trial results within 12 months of completion of the trial.